CLINICAL TRIAL: NCT00003390
Title: A Phase II Trial of 6-Hydroxymethylacylfulvene (MGI-114) in Patients With Advanced Renal Cell Carcinoma
Brief Title: 6-Hydroxymethylacylfulvene in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000066388; MSKCC-98009; MSKCC-98007; NCI-T97-0119
Record Dates: First submitted 1999-11-01; First posted 2004-08-26 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2000-05

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — irofulven

INTERVENTIONS:
Drug: irofulven

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of 6-hydroxymethylacylfulvene in treating patients with metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Evaluate the efficacy of 6-hydroxymethylacylfulvene (HMAF) in patients with metastatic renal cell carcinoma. II. Investigate the safety of HMAF given to this patient population.

OUTLINE: Patients receive 6-hydroxymethylacylfulvene intravenously for 5 minutes every day for 5 consecutive days. Treatment is repeated every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed after every 2 treatment courses.

PROJECTED ACCRUAL: Approximately 12-37 patients will be accrued for this study within 6-19 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed renal cell carcinoma and evidence of metastatic disease Bidimensionally measurable disease No active brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 70-100% Life expectancy: Greater than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin within normal range ALT/AST no greater than 2.5 times upper limit of normal (ULN) Renal: Creatinine within 1.5 times ULN AND Creatinine clearance at least 50 mL/min Other: Not pregnant or lactating Fertile patients must use effective contraception No prior malignancy within 5 years and at low risk for recurrence Must have undergone potentially curative therapy for prior malignancy

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since biological therapy and recovered Chemotherapy: No prior cytotoxic chemotherapy Endocrine therapy: At least 4 weeks since hormone therapy and recovered Radiotherapy: At least 4 weeks since radiotherapy Surgery: At least 4 weeks since major surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-06; Study Completion 2004-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Berg, MD, Study Chair — Sanofi
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States